CLINICAL TRIAL: NCT06051799
Title: Effects of Pressure Release of Myofascial Trigger Points on Mechanical Neck Pain. Randomised Controlled Clinical Trial.
Brief Title: Effects of Pressure Release of Myofascial Trigger Points on Mechanical Neck Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Iván Batuecas Sánchez, PhD student, Principal investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23/186-EC_X_Tesis
Record Dates: First submitted 2023-09-14; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Myofascial Pain Syndrome of Neck; Trigger Point Pain, Myofascial; Myofacial Pain
Keywords: upper trapezius; sternocleidomastoid; manual therapy; trigger points; Myofascial pain syndrome; therapeutic exercise
MeSH Terms: conditions — Myofascial Pain Syndromes; Facial Pain | interventions — Acupressure; Continuous Positive Airway Pressure; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, clinical trial with blinded assessment of response variables. The guidelines of the CONSORT guide will be followed.
  A follow-up of the participants will be carried out, where measurements will be taken prior to the intervention (baseline), after the protocol of four treatment sessions and fifteen days after the last session.
Who Masked: Participant, Outcomes Assessor
Masking Description: The selection of participants and the randomisation sequence will be carried out by the principal investigator using the patient's unique identity number in the centre's programme as a code. After randomisation, participants will be sent by another therapist in the centre to each intervention room without knowing which treatment they will receive. The therapists in charge of delivering the interventions will not know which patient has been assigned to them.
  Although both therapists and patients will not know which group they are assigned to, obviously the therapist, given the nature of the intervention and the need to know and master the technique, knows which treatment to apply to each subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TREATMENT GROUP (Experimental): The Pressure Release Technique will be applied. One session per week will be carried out for four weeks. It will be performed on as many trigger points as we find in each muscle associated with the study, leaving a record of them. Also adding postural hygiene and home exercise guidelines. A progression of exercises involving contraction of the deep neck flexor muscles Subjects will be taught to perform slow and controlled craniocervical flexion. It should be performed a minimum of once daily during the treatment regimen. A follow-up of the patients will be carried out with respect to home therapeutic exercise and postural hygiene guidelines.
  Interventions: Other: Myofascial trigger points pressure release; Other: Therapeutic exercise and postural hygiene
- CONTROL (Active Comparator): Postural hygiene guidelines will be given, as well as home therapeutic exercise (identical to the treatment group). About therapeutic exercise, a progression of exercises involving contraction of the deep neck flexor muscles shall be included in the first session. Subjects will be taught to perform slow and controlled craniocervical flexion. Subjects will then be trained to be able to progressively maintain craniocervical flexion through feedback from an air device (Stabilizer™, Chattanooga Group Inc., Chattanooga, TN) placed behind the neck. This sensor monitors the slight flattening of the cervical curve that occurs with contraction of the craniocervical deep flexor musculature. It should be performed a minimum of once daily during the treatment regimen. To this end, patients will be monitored and their understanding and correct follow-up of the treatment will be assessed in each face-to-face session per week, for four weeks, the same as in experimental group.
  Interventions: Other: Therapeutic exercise and postural hygiene

INTERVENTIONS:
Other: Myofascial trigger points pressure release — Patient lying down in the supine position, Therapist do a first and second finger pincer grasp is performed on the myofascial trigger points located on the upper trapezius muscle and sternocleidomastoid muscle, this pressure will be increased as the therapist perceives a reduction in soft tissue resistance under the finger over a period of 90 seconds. Previous studies indicate no difference between 60 and 90 seconds of pressure. It will be performed on as many trigger points as we find in each muscle associated with the study.
  Other Names: Ischemic compression; pressure release; manual compression
  Arms: TREATMENT GROUP
Other: Therapeutic exercise and postural hygiene — Therapeutic exercise and postural hygiene: A progression of exercises with contraction of the deep neck flexor muscles will be included in the first session. Subjects will be taught to perform a slow and controlled craniocervical flexion. Subjects will then be trained to be able to progressively maintain craniocervical flexion through feedback from an air device (Stabilizer™, Chattanooga Group Inc., Chattanooga, TN) placed behind the neck. This sensor monitors the slight flattening of the cervical curve that occurs with contraction of the craniocervical deep flexor musculature. It should be performed at least once a day during the treatment regimen.
  Also Postural correction exercises carried out regularly throughout the day, especially when seated. Indications are given to avoid pelvic retroversion and maintain a natural lumbar lordosis while performing retraction and adduction of the scapulae and gently lengthening the spine.
  Other Names: postural correction; motor control exercise

SUMMARY:
The study aims to compare the effectiveness of myofascial trigger point treatment using pressure release versus a control group in patients with mechanical neck pain, randomly assigned. In both groups a protocol of therapeutic exercise and postural correction will be carried out

DETAILED DESCRIPTION:
With the present investigation it is wondered whether the choice of manual therapy techniques, specifically the pressure release of myofascial trigger points in the upper trapezius and sternocleidomastoid muscles, provide significant benefits in combination with therapeutic exercise and postural hygiene (treatment group), as opposed to the unique application of therapeutic exercise and postural hygiene (control group), thus constituting a treatment of choice in patients with mechanical neck pain.

A treatment protocol of one session per week will be carried out, and a follow-up two weeks after the end of the treatment protocol.

If, as postulated, pressure release is more effective than the treatment received by the control group, the choice of this type of technique for myofascial pain syndrome would benefit a high percentage of people who often come asking for treatment in pain treatment centers. Pressure release provides a painless manual stimulus, thus effectively resolving the symptomatology of myofascial trigger points without the need for invasive treatments or medication, which may have more contraindications.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 55 years of age in order to avoid degenerative phenomena.
* Have suffered from neck pain at least once in the last month.
* Active or latent myofascial trigger points in the Upper Trapezius and Sternocleidomastoid muscles.

Exclusion Criteria:

* Patients with recent trauma (last 6 months) to the upper quadrant or spine.
* Patients with pathologies involving malignant neoplasms.
* Surgery on the trunk or upper limb in the last six months.
* Patients undergoing pharmacological or physiotherapy treatment at the time of the test.
* Pregnancy.
* No myofascial trigger points in the upper trapezius or sternocleidomastoid muscles.
* Refusal to sign the consent form for the study or not being able to do so.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-09-25 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale. Base | Baseline. Prior to the first treatment session
  Measure of pain intensity. A mark is placed on a 10-centimetre line with the left end being no pain at all and the right end being the worst pain imaginable.
Visual analogue scale. Post treatment | Up to 4 weeks. After the end protocol of four treatment sessions
  Measure of pain intensity. A mark is placed on a 10-centimetre line with the left end being no pain at all and the right end being the worst pain imaginable.
Visual analogue scale. Follow up | Follow-up two weeks after the end of the four-session treatment protocol
  Measure of pain intensity. A mark is placed on a 10-centimetre line with the left end being no pain at all and the right end being the worst pain imaginable.
Pressure pain threshold. Base | Baseline. Prior to the first treatment session
  Measurement of pain threshold to pressure with Fischer algometer. The algometer is placed perpendicular to the myofascial trigger point previously marked by the therapist. Once in place, the pressure is increased at a rate of 1 kilogram per second (kg per sec) until the patient begins to feel discomfort. At this point, the application is stopped. Three measurements are taken and the average is calculated.
Pressure pain threshold. Post treatment | Up to 4 weeks. After the end protocol of four treatment sessions
  Measurement of pain threshold to pressure with Fischer algometer. The algometer is placed perpendicular to the myofascial trigger point previously marked by the therapist. Once in place, the pressure is increased at a rate of 1 kilogram per second (kg per sec) until the patient begins to feel discomfort. At this point, the application is stopped. Three measurements are taken and the average is calculated.
Pressure pain threshold. Follow up | Follow-up two weeks after the end of the four-session treatment protocol
  Measurement of pain threshold to pressure with Fischer algometer. The algometer is placed perpendicular to the myofascial trigger point previously marked by the therapist. Once in place, the pressure is increased at a rate of 1 kilogram per second (kg per sec) until the patient begins to feel discomfort. At this point, the application is stopped. Three measurements are taken and the average is calculated.
Cervical Disability Index. Base | Baseline. Prior to the first treatment session
  Results on the Northwick Park Cervical Spine Disability Questionnaire, translated and validated in Spanish. The pre-questionnaire consists of 9 questions related to pain intensity, sleep, weight bearing, leisure and social activities, work and driving. Each question has 5 possible answers ranging from 0 to 4, where 0 represents the absence of disability and 4 the maximum degree of disability. Similarly, the subsequent questionnaire consists of 10 questions and the same answers. Taking this into account, the maximum score that can be obtained would be 36 in the pre-questionnaire or 40 in the post-questionnaire (categorised as high disability).
Cervical Disability Index. Post treatment | Up to 4 weeks. After the end protocol of four treatment sessions
  Results on the Northwick Park Cervical Spine Disability Questionnaire, translated and validated in Spanish. The pre-questionnaire consists of 9 questions related to pain intensity, sleep, weight bearing, leisure and social activities, work and driving. Each question has 5 possible answers ranging from 0 to 4, where 0 represents the absence of disability and 4 the maximum degree of disability. Similarly, the subsequent questionnaire consists of 10 questions and the same answers. Taking this into account, the maximum score that can be obtained would be 36 in the pre-questionnaire or 40 in the post-questionnaire (categorised as high disability).
Cervical Disability Index. Follow up | Follow-up two weeks after the end of the four-session treatment protocol
  Results on the Northwick Park Cervical Spine Disability Questionnaire, translated and validated in Spanish. The pre-questionnaire consists of 9 questions related to pain intensity, sleep, weight bearing, leisure and social activities, work and driving. Each question has 5 possible answers ranging from 0 to 4, where 0 represents the absence of disability and 4 the maximum degree of disability. Similarly, the subsequent questionnaire consists of 10 questions and the same answers. Taking this into account, the maximum score that can be obtained would be 36 in the pre-questionnaire or 40 in the post-questionnaire (categorised as high disability).
Pain catastrophising scale. Base | Baseline. Prior to the first treatment session.
  It is the set of cognitive and emotional processes consisting of having negative thoughts about the future that predispose to the chronification of pain. Self-administered scale made up of 13 items, each item scored from 0 to 4. The total score range is from 0 to 52, where higher scores indicate a higher level of catastrophism. It is one of the most widely used to assess the pain catastrophising construct.
Pain catastrophising scale. Post treatment | Up to 4 weeks. After the end protocol of four treatment sessions
  It is the set of cognitive and emotional processes consisting of having negative thoughts about the future that predispose to the chronification of pain. Self-administered scale made up of 13 items, each item scored from 0 to 4. The total score range is from 0 to 52, where higher scores indicate a higher level of catastrophism. It is one of the most widely used to assess the pain catastrophising construct.
Pain catastrophising scale. Follow up | Follow-up two weeks after the end of the four-session treatment protocol
  It is the set of cognitive and emotional processes consisting of having negative thoughts about the future that predispose to the chronification of pain. Self-administered scale made up of 13 items, each item scored from 0 to 4. The total score range is from 0 to 52, where higher scores indicate a higher level of catastrophism. It is one of the most widely used to assess the pain catastrophising construct.
Tampa Kinesiophobia Scale (ETK-11). Base | Baseline. Prior to the first treatment session.
  Translated into Spanish. It is one of the most frequently used measures to assess pain-related fear of movement in patients with chronic pain. The ETK-11 is an 11-item self-questionnaire in its Spanish version that measures fear of movement and pain. The total score of the ETK-11 is between 11 - 44 points and each item has a likert scale that scores from 1 to 4 (1 = strongly disagree, 4 = strongly agree). Higher scores indicate greater fear of movement and pain. The ETK-11 has two subscales: activity avoidance and harm avoidance.
Tampa Kinesiophobia Scale (ETK-11). Post treatment | Up to 4 weeks. After the end protocol of four treatment sessions
  Translated into Spanish. It is one of the most frequently used measures to assess pain-related fear of movement in patients with chronic pain. The ETK-11 is an 11-item self-questionnaire in its Spanish version that measures fear of movement and pain. The total score of the ETK-11 is between 11 - 44 points and each item has a likert scale that scores from 1 to 4 (1 = strongly disagree, 4 = strongly agree). Higher scores indicate greater fear of movement and pain. The ETK-11 has two subscales: activity avoidance and harm avoidance.
Tampa Kinesiophobia Scale (ETK-11). Follow up | Follow-up two weeks after the end of the four-session treatment protocol
  Translated into Spanish. It is one of the most frequently used measures to assess pain-related fear of movement in patients with chronic pain. The ETK-11 is an 11-item self-questionnaire in its Spanish version that measures fear of movement and pain. The total score of the ETK-11 is between 11 - 44 points and each item has a likert scale that scores from 1 to 4 (1 = strongly disagree, 4 = strongly agree). Higher scores indicate greater fear of movement and pain. The ETK-11 has two subscales: activity avoidance and harm avoidance.

SECONDARY OUTCOMES:
Swallow-wall distance. Base | Baseline. Prior to the first treatment session.
  Patient in a sitting position, back against the wall, the distance in centimetres is measured using a tape measure or ruler between the swallow and the surface of the wall during the maximum effort to bring the head close to the wall. The chin should not be lifted higher than horizontal. The average of both sides gives the final result. A value greater than 15 centimetres is considered pathological.
Swallow-wall distance. Post treatment | Up to 4 weeks. After the end protocol of four treatment sessions
  Patient in a sitting position, back against the wall, the distance in centimetres is measured using a tape measure or ruler between the swallow and the surface of the wall during the maximum effort to bring the head close to the wall. The chin should not be lifted higher than horizontal. The average of both sides gives the final result. A value greater than 15 centimetres is considered pathological.
Swallow-wall distance. Follow up | Follow-up two weeks after the end of the four-session treatment protocol
  Patient in a sitting position, back against the wall, the distance in centimetres is measured using a tape measure or ruler between the swallow and the surface of the wall during the maximum effort to bring the head close to the wall. The chin should not be lifted higher than horizontal. The average of both sides gives the final result. A value greater than 15 centimetres is considered pathological.
Cervical flexion-extension. Base | Baseline. Prior to the first treatment session.
  Using the "Goniometer pro" mobile app. The patient performs flexion and extension movements and the inclinometer of the mobile device records the degrees of movement. Three measurements are taken and the average is recorded.
Cervical flexion-extension. Post treatment | Up to 4 weeks. After the end protocol of four treatment sessions.
  Using the "Goniometer pro" mobile app. The patient performs flexion and extension movements and the inclinometer of the mobile device records the degrees of movement. Three measurements are taken and the average is recorded.
Cervical flexion-extension. Follow up | Follow-up two weeks after the end of the four-session treatment protocol.
  Using the "Goniometer pro" mobile app. The patient performs flexion and extension movements and the inclinometer of the mobile device records the degrees of movement. Three measurements are taken and the average is recorded.
Cervical rotation. Base | BaselinePrior to the first treatment session.
  Via mobile application "Goniometer pro". The patient performs a cervical rotation movement to the left and right side and the degrees of movement are recorded by recording the angular translation of the mobile device on the apex of the skull. Three measurements are taken and the mean is recorded.
Cervical rotation. Post treatment | Up to 4 weeks. After the end protocol of four treatment sessions.
  Via mobile application "Goniometer pro". The patient performs a cervical rotation movement to the left and right side and the degrees of movement are recorded by recording the angular translation of the mobile device on the apex of the skull. Three measurements are taken and the mean is recorded.
Cervical rotation. Follow up | Follow-up two weeks after the end of the four-session treatment protocol.
  Via mobile application "Goniometer pro". The patient performs a cervical rotation movement to the left and right side and the degrees of movement are recorded by recording the angular translation of the mobile device on the apex of the skull. Three measurements are taken and the mean is recorded.
Side bending. Base | Baseline. Prior to the first treatment session.
  Using the "Goniometer pro" mobile app. The patient performs a lateral tilt movement to the right and left side and the degrees of movement are recorded using the inclinometer on the mobile device. The device is placed vertically on the prominence of the spinous process of the 7th cervical vertebra following the tilt movement. Three measurements shall be taken and the mean shall be recorded.
Side bending. Post treatment | Up to 4 weeks. After the end protocol of four treatment sessions.
  Using the "Goniometer pro" mobile app. The patient performs a lateral tilt movement to the right and left side and the degrees of movement are recorded using the inclinometer on the mobile device. The device is placed vertically on the prominence of the spinous process of the 7th cervical vertebra following the tilt movement. Three measurements shall be taken and the mean shall be recorded.
Side bending. Follow up | Follow-up two weeks after the end of the four-session treatment protocol.
  Using the "Goniometer pro" mobile app. The patient performs a lateral tilt movement to the right and left side and the degrees of movement are recorded using the inclinometer on the mobile device. The device is placed vertically on the prominence of the spinous process of the 7th cervical vertebra following the tilt movement. Three measurements shall be taken and the mean shall be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Angela C Álvarez Melcón, Doctor, Study Director — Universidad Complutense de Madrid; Isidro Fernández López, Doctor, Study Director — Universidad Complutense de Madrid; María A Atín Arratibel, Doctor, Study Director — Universidad Complutense de Madrid; Iván Batuecas Sánchez, PhD, Principal Investigator — Universidad Complutense / Fisioterapia Los Molinos
Locations (1):
- Fisioterapia Los Molinos, Getafe, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The present study is carried out as a doctoral thesis of the principal investigator. Therefore, a scientific dissemination is foreseen in the Complutense University of Madrid as well as in the appropriate journals.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From July 2024 until the submission of the thesis
Access Criteria: Upon request to the principal investigator and his research team

REFERENCES:
- [Result] Munoz-Munoz S, Munoz-Garcia MT, Alburquerque-Sendin F, Arroyo-Morales M, Fernandez-de-las-Penas C. Myofascial trigger points, pain, disability, and sleep quality in individuals with mechanical neck pain. J Manipulative Physiol Ther. 2012 Oct;35(8):608-13. doi: 10.1016/j.jmpt.2012.09.003. PMID 23158466
- [Result] Cerezo-Tellez E, Torres-Lacomba M, Mayoral-Del Moral O, Sanchez-Sanchez B, Dommerholt J, Gutierrez-Ortega C. Prevalence of Myofascial Pain Syndrome in Chronic Non-Specific Neck Pain: A Population-Based Cross-Sectional Descriptive Study. Pain Med. 2016 Dec;17(12):2369-2377. doi: 10.1093/pm/pnw114. Epub 2016 Jun 20. PMID 28025371
- [Result] Chao YW, Lin JJ, Yang JL, Wang WT. Kinesio taping and manual pressure release: Short-term effects in subjects with myofasical trigger point. J Hand Ther. 2016 Jan-Mar;29(1):23-9. doi: 10.1016/j.jht.2015.10.003. Epub 2015 Nov 6. PMID 26705672
- [Result] Grieve R, Barnett S, Coghill N, Cramp F. The prevalence of latent myofascial trigger points and diagnostic criteria of the triceps surae and upper trapezius: a cross sectional study. Physiotherapy. 2013 Dec;99(4):278-84. doi: 10.1016/j.physio.2013.04.002. Epub 2013 Jul 2. PMID 23830716
- [Result] Oliveira-Campelo NM, de Melo CA, Alburquerque-Sendin F, Machado JP. Short- and medium-term effects of manual therapy on cervical active range of motion and pressure pain sensitivity in latent myofascial pain of the upper trapezius muscle: a randomized controlled trial. J Manipulative Physiol Ther. 2013 Jun;36(5):300-9. doi: 10.1016/j.jmpt.2013.04.008. Epub 2013 Jun 12. PMID 23769263
- [Result] Cagnie B, Castelein B, Pollie F, Steelant L, Verhoeyen H, Cools A. Evidence for the Use of Ischemic Compression and Dry Needling in the Management of Trigger Points of the Upper Trapezius in Patients with Neck Pain: A Systematic Review. Am J Phys Med Rehabil. 2015 Jul;94(7):573-83. doi: 10.1097/PHM.0000000000000266. PMID 25768071
- [Result] De Meulemeester KE, Castelein B, Coppieters I, Barbe T, Cools A, Cagnie B. Comparing Trigger Point Dry Needling and Manual Pressure Technique for the Management of Myofascial Neck/Shoulder Pain: A Randomized Clinical Trial. J Manipulative Physiol Ther. 2017 Jan;40(1):11-20. doi: 10.1016/j.jmpt.2016.10.008. PMID 28017188
- [Result] Pecos-Martin D, Ponce-Castro MJ, Jimenez-Rejano JJ, Nunez-Nagy S, Calvo-Lobo C, Gallego-Izquierdo T. Immediate effects of variable durations of pressure release technique on latent myofascial trigger points of the levator scapulae: a double-blinded randomised clinical trial. Acupunct Med. 2019 Jun;37(3):141-150. doi: 10.1136/acupmed-2018-011738. Epub 2019 May 7. PMID 31060367
- [Result] Fernandez-de-Las-Penas C, Dommerholt J. International Consensus on Diagnostic Criteria and Clinical Considerations of Myofascial Trigger Points: A Delphi Study. Pain Med. 2018 Jan 1;19(1):142-150. doi: 10.1093/pm/pnx207. PMID 29025044
- [Result] Tsiringakis G, Dimitriadis Z, Triantafylloy E, McLean S. Motor control training of deep neck flexors with pressure biofeedback improves pain and disability in patients with neck pain: A systematic review and meta-analysis. Musculoskelet Sci Pract. 2020 Dec;50:102220. doi: 10.1016/j.msksp.2020.102220. Epub 2020 Jul 24. PMID 32827852
- [Result] de Zoete RM, Armfield NR, McAuley JH, Chen K, Sterling M. Comparative effectiveness of physical exercise interventions for chronic non-specific neck pain: a systematic review with network meta-analysis of 40 randomised controlled trials. Br J Sports Med. 2020 Nov 2:bjsports-2020-102664. doi: 10.1136/bjsports-2020-102664. Online ahead of print. PMID 33139256
- [Result] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; CONSORT. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2012;10(1):28-55. doi: 10.1016/j.ijsu.2011.10.001. Epub 2011 Oct 12. PMID 22036893
- [Result] Hou CR, Tsai LC, Cheng KF, Chung KC, Hong CZ. Immediate effects of various physical therapeutic modalities on cervical myofascial pain and trigger-point sensitivity. Arch Phys Med Rehabil. 2002 Oct;83(10):1406-14. doi: 10.1053/apmr.2002.34834. PMID 12370877
- [Result] Jull GA, O'Leary SP, Falla DL. Clinical assessment of the deep cervical flexor muscles: the craniocervical flexion test. J Manipulative Physiol Ther. 2008 Sep;31(7):525-33. doi: 10.1016/j.jmpt.2008.08.003. PMID 18804003
- [Result] Rodriguez-Sanz J, Malo-Urries M, Corral-de-Toro J, Lopez-de-Celis C, Lucha-Lopez MO, Tricas-Moreno JM, Lorente AI, Hidalgo-Garcia C. Does the Addition of Manual Therapy Approach to a Cervical Exercise Program Improve Clinical Outcomes for Patients with Chronic Neck Pain in Short- and Mid-Term? A Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Sep 10;17(18):6601. doi: 10.3390/ijerph17186601. PMID 32927858
- [Result] Tsang SMH, So BCL, Lau RWL, Dai J, Szeto GPY. Effects of combining ergonomic interventions and motor control exercises on muscle activity and kinematics in people with work-related neck-shoulder pain. Eur J Appl Physiol. 2018 Apr;118(4):751-765. doi: 10.1007/s00421-018-3802-6. Epub 2018 Jan 15. PMID 29335773
- [Result] Beer A, Treleaven J, Jull G. Can a functional postural exercise improve performance in the cranio-cervical flexion test?--a preliminary study. Man Ther. 2012 Jun;17(3):219-24. doi: 10.1016/j.math.2011.12.005. Epub 2012 Feb 4. PMID 22310655
- [Result] Boonstra AM, Schiphorst Preuper HR, Balk GA, Stewart RE. Cut-off points for mild, moderate, and severe pain on the visual analogue scale for pain in patients with chronic musculoskeletal pain. Pain. 2014 Dec;155(12):2545-2550. doi: 10.1016/j.pain.2014.09.014. Epub 2014 Sep 17. PMID 25239073
- [Result] Park G, Kim CW, Park SB, Kim MJ, Jang SH. Reliability and usefulness of the pressure pain threshold measurement in patients with myofascial pain. Ann Rehabil Med. 2011 Jun;35(3):412-7. doi: 10.5535/arm.2011.35.3.412. Epub 2011 Jun 30. PMID 22506152
- [Result] Gonzalez T, Balsa A, Sainz de Murieta J, Zamorano E, Gonzalez I, Martin-Mola E. Spanish version of the Northwick Park Neck Pain Questionnaire: reliability and validity. Clin Exp Rheumatol. 2001 Jan-Feb;19(1):41-6. PMID 11247324
- [Result] Garcia Campayo J, Rodero B, Alda M, Sobradiel N, Montero J, Moreno S. [Validation of the Spanish version of the Pain Catastrophizing Scale in fibromyalgia]. Med Clin (Barc). 2008 Oct 18;131(13):487-92. doi: 10.1157/13127277. Spanish. PMID 19007576
- [Result] Gomez-Perez L, Lopez-Martinez AE, Ruiz-Parraga GT. Psychometric Properties of the Spanish Version of the Tampa Scale for Kinesiophobia (TSK). J Pain. 2011 Apr;12(4):425-35. doi: 10.1016/j.jpain.2010.08.004. PMID 20926355
- [Result] Vohralik SL, Bowen AR, Burns J, Hiller CE, Nightingale EJ. Reliability and validity of a smartphone app to measure joint range. Am J Phys Med Rehabil. 2015 Apr;94(4):325-30. doi: 10.1097/PHM.0000000000000221. PMID 25299533
- [Result] Melian-Ortiz A, Varillas-Delgado D, Laguarta-Val S, Rodriguez-Aparicio I, Senent-Sansegundo N, Fernandez-Garcia M, Roger-de Ona I. [Reliability and concurrent validity of the app Goniometer Pro vs Universal Goniometer in the determination of passive knee flexion]. Acta Ortop Mex. 2019 Jan-Feb;33(1):18-23. Spanish. PMID 31480121
- [Result] Ghorbani F, Kamyab M, Azadinia F. Smartphone Applications as a Suitable Alternative to CROM Device and Inclinometers in Assessing the Cervical Range of Motion in Patients With Nonspecific Neck Pain. J Chiropr Med. 2020 Mar;19(1):38-48. doi: 10.1016/j.jcm.2019.10.004. Epub 2020 Sep 3. PMID 33192190
- [Result] Pourahmadi MR, Bagheri R, Taghipour M, Takamjani IE, Sarrafzadeh J, Mohseni-Bandpei MA. A new iPhone application for measuring active craniocervical range of motion in patients with non-specific neck pain: a reliability and validity study. Spine J. 2018 Mar;18(3):447-457. doi: 10.1016/j.spinee.2017.08.229. Epub 2017 Sep 7. PMID 28890223